CLINICAL TRIAL: NCT05282394
Title: Newborn Abdominal Massage to Prevent Hyperbilirubinemia: A Pilot Randomized Controlled Trial
Brief Title: Newborn Abdominal Massage to Prevent Hyperbilirubinemia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1817729; K12HD051958 (NIH)
Record Dates: First submitted 2021-12-14; First posted 2022-03-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Newborn Jaundice
Keywords: newborn massage
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage Intervention (Experimental): Families will be instructed to provide parent-provided newborn abdominal massage three times per day through 5 days of life
  Interventions: Procedure: Abdominal massage
- Attention Control Intervention (Other): Families will be provided with information about reading with baby.
  Interventions: Other: Reading

INTERVENTIONS:
Procedure: Abdominal massage — abdominal massage
  Arms: Massage Intervention
Other: Reading — guidance given to parents about reading with baby
  Arms: Attention Control Intervention

SUMMARY:
The proposed study will incorporate an intervention previously un-studied in the US healthcare setting for prevention of hyperbilirubinemia

ELIGIBILITY:
Inclusion Criteria:

* Newborn admitted to the well newborn/postpartum care unit at UC Davis Medical Center
* Less than 48 hours of age at enrollment

Exclusion Criteria:

* Infant has already received phototherapy
* Mother/birthing person is incarcerated
* Infant unexpected to discharge into parental care
* Parental inability to speak or read in English
* Infant without parent rooming-in with them in the hospital

Ages: 0 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the newborn massage intervention | Through study completion, up to one year
  Acceptability of the intervention will be defined by the 1-sided 95% confidence interval for the proportion of the intervention group performing massage at least once to include 80% and for the 1-sided 95% confidence interval for at the proportion performing massage as directed to include 70%.
Feasibility of recruitment | Ascertained following completion of recruitment of 30 study participants. Through study completion, up to an average of one year.
  Feasibility of recruitment will be defined by at least 30% of approached, eligible participants consenting to participate.

SECONDARY OUTCOMES:
Difference between transcutaneous bilirubin level and AAP phototherapy threshold on the day of discharge | Value at obtained at hospital discharge will be evaluated at the end of study completion, up to one year
  delta-TcSB, which is calculated by subtracting infant's transcutaneous bilirubin level from their phototherapy treatment threshold at that hour of age (in mg/dL)
Number of stools in prior 24 hours (at hospital discharge) | Value at obtained at hospital discharge will be evaluated at the end of study completion, up to one year
Timing of first transitional (non-meconium) stool passage | Ascertained at 1-2 week survey
Parental satisfaction with newborn massage | 7-14 day survey
  Parental satisfaction with newborn massage assessed by survey
Proportion of participants who read with baby in the last 24 hours | 1-2 week survey
  Proportion of participants who read with baby in the last 24 hours assessed by survey
Proportion of participants who read with baby in the last week | 1-2 week survey
  Proportion of participants who read with baby in the last week assessed by survey
Breastfeeding at 1 week of age | 1-2 week survey
  Infant received any human milk in the prior 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kair, MD, MAS, Principal Investigator — UC Davis Health
Locations (1):
- University of California-Davis, Sacramento, California, United States